CLINICAL TRIAL: NCT01097564
Title: COL4A1 Gene Related Cerebra-retinal Angiopathy : Clinical Spectrum From Children to Adult, Mutational Spectrum and Application to Routine Management of Affected Patients : a Prospective Cohort Study
Brief Title: COL4A1 Gene Related Cerebra-retinal Angiopathy
Acronym: COL4A1
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P081214; 2009-A01163-54 (Other: IDRCB)
Record Dates: First submitted 2010-02-19; First posted 2010-04-01 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Cerebra-retinal Angiopathy
Keywords: Genetic; Cerebral angiopathy; Retinal angiopathy; COL4A1 gene; Infantile Cerebral Palsy; Congenital porencephaly; Congenital cataract; Leukoencephalopathy; COL4A1 gene related cerebra-retinal angiopathy
MeSH Terms: conditions — Cerebral Palsy; Porencephaly; Leukoencephalopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COL4A1 genetic testing: COL4A1 genetic testing
  Interventions: Genetic: COL4A1 genetic testing

INTERVENTIONS:
Genetic: COL4A1 genetic testing — genetic testing

SUMMARY:
This prospective multicenter cohort study aims to define the clinical, radiological and mutational spectrum of the disease related to COL4A1 gene.

DETAILED DESCRIPTION:
150 index patients (children or young adult) will be prospectively recruited over three years according to eligibility criteria. Relatives will be also recruited.

Clinical, brain MRI-MRA and genetic testing (COL4A1 mutation screening) will be conducted for each included patient or asymptomatic relatives. 13 French investigating centres will be participating to the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the index patient :

* Children and young adult (< 65 years)
* Intracranial hemorrhage of unknown etiology
* leukoencephalopathy
* Any associated signs (including retinal arteriolar tortuosity, intracranial aneurysm, porencephaly, Infantile Cerebral Palsy, juvenile cataract)

Exclusion criteria:

(for the index patient)

* Hypertension
* Diabetes
* Other (than COL4A1) genetic small vessel diseases of the brain

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * patients children
  * patients young adult
  * family adult symptomatic
  * family adult asymptomatic
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2010-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Implication of COL4A1 gene (and other related genes) in intracranial haemorrhages of unknown etiology in children and young adults and in brain diffuse small vessel diseases of unknown etiology in young adults. | at 36 months

SECONDARY OUTCOMES:
To define the whole clinical, radiological and mutational spectrum of COL4A1 gene. | at 36 months
To define any genotype-phenotype correlation in COL4A1 gene disease. | at 36 months
Application of the results in daily clinical practice | at 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugues CHABRIAT, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital LARIBOISIERE Neurology Department, Paris, France